CLINICAL TRIAL: NCT02374008
Title: The Effect of Saphenous Nerve and Obturator Nerve Block Combined With Systemic High Dose Glucocorticoid Versus Local Infiltration Analgesia Combined With a Systemic High Dose Glucocorticoid on Opioid Consumption and Pain After Total Knee Arthroplasty
Brief Title: The Analgesic Effect of Combined Nerve Block and Systemic High Dose Glucocorticoid After Total Knee Arthroplasty.
Acronym: HOBSALIplus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Silkeborg (Other)
Responsible Party: Principal Investigator, Charlotte Runge, MD, Ph.D student, Regionshospitalet Silkeborg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-003343-35
Record Dates: First submitted 2015-02-22; First posted 2015-02-27 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Peripheral Nerve Block; Pain
Keywords: Peripheral nerve block; Total knee Arthroplasty; Dexamethasone
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Epinephrine; Ketorolac; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined nerve block (Experimental): Ropivacaine and Adrenalin, systemic Ketorolac and high dose Dexamethasone
  Interventions: Drug: Ropivacaine
- Local infiltrationanalgesia (Active Comparator): Ropivacaine, Adrenalin and Ketorolac combined with systemic high dose dexamethasone
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine
  Other Names: Adrenalin; Ketorolac; Dexamethasone

SUMMARY:
Purpose:

The purpose of this study is to evaluate the postoperative analgesic effect of a combined Saphenous nerve block and Obturator nerve block with local infiltration analgesia in the tissue around the knee after total kneearthroplasty. In the combined nerve blocks we use a mixture of Ropivacaine and Adrenaline combined with high dose systemic dexamethasone and Ketorolac and the mixture for local infiltration consist of Ropivacaine, Adrenaline and Ketoroloc. The investigators hypothesis is that the combined nerve blocks reduces pain and reduces the opioid consumption and thus reduce side effects such as nausea, vomiting and lethargy compared to the current treatment with local infiltration analgesia.

Background:

Nerve blocks as analgesic treatment after orthopedic surgery is a recognized and proven procedure. The nerve blocks have the disadvantage that not only do they anesthetize the sensory nerve fibers but also the nerve fibers to the muscles of the leg. The Saphenous nerve block causes only stunning of sensory nerves to the knee region. The Obturator nerve block causes both stunning of the sensory nerves to the knee region and the thighs inward leading muscles, and does not affect the patient's mobilization capacity.

Both blocks are known to be a good addition to the analgesic treatment. Ropivacaine is a well-known local anesthetic. Adrenaline have also been used in other studies, in addition to the local anesthetic agent, and has been shown to prolong the effect of the nerve block. Saphenous and Obturator nerve block with all four drugs Ropivacaine and Adrenaline combined with high dose systemic Dexamethasone has not been systematically investigated in knee replacement surgery, and it is not known whether this method will provide better pain treatment.

Method

The patient can receive one of two treatments, determined randomly:

* A. Saphenous and Obturator nerve block with active anesthetics (Ropivacaine, Adrenaline) combined with systemic ketoroloc and high dose Dexamethasone and local infiltration around the knee joint with placebo medicine (normal saline).
* B. Both blocks with placebo medicine (normal saline) and local infiltration around the knee joint with activ local anesthetic.

Neither patient, investigator or staff around the patient will have knowledge of which treatment the patient has received.

The blocks will be placed before the operation and local infiltration around the knee joint will be given by the surgeon during the operation.

ELIGIBILITY:
Inclusion Criteria:

* Age> 50 years
* Patients set to cemented Total knee arthroplasty in spinal block
* ASA 1-3

Exclusion Criteria:

* Patients who can not cooperate with the investigation
* Patients who have given written informed consent to participate in the study after having understood the contents of the protocol and limitations fully
* Patients who do not understand or speak Danish
* Patients receiving immunosuppressive therapy
* Patients receiving glucocorticoid daily
* Patients with a treatment-dependent diabetes mellitus
* Patients with known neuropathy in the lower limbs
* Allergy to those used in the study drugs
* Alcohol and / or drug abuse - the investigator's opinion
* Patients who can not tolerate NSAIDs
* Fixed several times daily consumption of strong opioids (morphine, ketogan, Oxynorm, methadone, fentanyl)

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 0 - 20 hours postoperatively

SECONDARY OUTCOMES:
Opioid consumption | 0 - 24 hours postoperatively
Pain Score by passive flexion of the knee joint from 0-90 degrees. | At timepoint 2 , 6, 20 and 24 hours postoperatively
  Using NRS (numeric rating scale) values from 0 to 10, with 0 being no pain and 10 being the worst pain imaginable.
Pain score at rest | At timepoint 2 , 6, 20 and 24 hours postoperatively
  Using NRS (numeric rating scale) values from 0 to 10, with 0 being no pain and 10 being the worst pain imaginable. The highest score since last score recorded.
Time of initial postoperative opioid-required pain breakthrough ( NRS > 3 at rest) | 0-24 hours postoperatively
  Recorded at PCA(patient-controlled-analgesia) pump
Nausea Score | At timepoint 2, 6, 20, 24 hours postoperatively
  NRS (numeric rating scale ) - with values from 0 to 10, where 0 is no nausea and 10 being the worst nausea. The highest score since last score recorded.
Number of vomiting | 0- 20 hours and 0-24 hours postoperatively
Consumption of Ondansetron | 0-20 hours and 0-24 hours
Reporting of dizziness Recording whether the dizziness is preventing mobilization. | at timepoint 2, 6, 20 and 24 hours postoperatively.
  Recording whether the dizziness is preventing
Duration of stay (length of stay , LOS ) in the observation unit (post anesthesia care unit , pacu). | 0-24 hours postoperatively
  The end time for the LOS in PACU recorded at the time when the patient meets DASAIMs (Danish Society of Anaesthesiology and Intensive Therapy) printing criteria - regardless of Pacu 's logistics in general.
Discharge time from the hospital | maximum 60 hour postoperatively.
Preoperatively isometric tests of muscle strength in the hip adductors. | pre and 30 minutes after block placement
  Performed by a handheld dynamometer before and 30 minutes after performed nerve blockades. The patient performed 4-10 measurements with a 30 second break in between each measurement. The difference between the highest value for the test before and after nerve block is calculated.
Time where the patient first time are mobilize to walk postoperatively with crutches or support from nurses. | 0-24 hours posteratively

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Runge, MD, Study Director — Regionalhospital Silkeborg

REFERENCES:
- [Derived] Runge C, Jensen JM, Clemmesen L, Knudsen HB, Holm C, Borglum J, Bendtsen TF. Analgesia of Combined Femoral Triangle and Obturator Nerve Blockade Is Superior to Local Infiltration Analgesia After Total Knee Arthroplasty With High-Dose Intravenous Dexamethasone. Reg Anesth Pain Med. 2018 May;43(4):352-356. doi: 10.1097/AAP.0000000000000731. PMID 29346228